CLINICAL TRIAL: NCT03714516
Title: LIVIA-FR: Non-controlled Evaluation of a French Unguided Internet-based Self-help Intervention for Adults Struggling With Prolonged Grief Symptoms After the Loss of Their Romantic Partner (Bereavement or Separation/Divorce)
Brief Title: Evaluation of a French Unguided Internet-based Intervention for Adults Struggling With Their Partner's Loss
Acronym: LIVIA-FR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne (Other)
Responsible Party: Principal Investigator, Debrot Anik, Principal Investigator, University of Lausanne
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018-00401
Record Dates: First submitted 2018-09-21; First posted 2018-10-22 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Complicated Grief

STUDY DESIGN:
Intervention Model Description: non-controlled evaluation pilot study with pre-, post- and follow-up assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online psychological intervention (Experimental): The intervention is a non-controlled unguided internet-based self-help intervention for adults who seek support for coping with prolonged grief symptoms after romantic bereavement or separation/ divorce. The self-help program consists of 10 text-based sessions based on cognitive-behavioral psychotherapy techniques.
  Interventions: Behavioral: Psychological internet intervention

INTERVENTIONS:
Behavioral: Psychological internet intervention — The intervention is a non-controlled unguided internet-based self-help intervention for adults who seek support for coping with prolonged grief symptoms after romantic bereavement or separation/ divorce. The self-help program consists of 10 text-based sessions based on cognitive-behavioral psychotherapy techniques.

SUMMARY:
The purpose of this study is to demonstrate the effectiveness of an unguided self-help program for people struggling with the loss of their partner, either by separation/divorce or death. The self-support program lasts 2 months and a half to 3 months. It was developed in German by a team from the University of Bern and has already proven its effectiveness. All participants will have direct access to the program (there will be no control group). The results obtained will be compared to those collected by the authors of the original program who administered the same intervention to a German-speaking population, however with support by e-mail.

Participation is open to anyone aged 20 or over who has lost their partner through bereavement, divorce or separation at least 6 months ago, and who has difficulty overcoming this loss. However, it is not possible to participate if the person is on psychotherapeutic therapy, has started or changed psychotropic medication or if the person has any risk of suicide. Alternative possibilities of treatment will be proposed.

The self-support consists of 10 modules, which contain information about the process of loss, self-reflection tasks, activities, questionnaires and self-observation grids. Participants are free to do the modules as many times as they wish. They will also be asked three times to complete questionnaires taking an average of 40 minutes. This will take place before the start of the program, at the end of the program, and 3 months after the end of the intervention.

At the end of the program, participants will be asked for feedback on the program. These data and remarks will allow to rethink and improve the care of people with difficulties overcoming the loss of a loved one.

Participants will be recruited by contacting various associations dealing with bereavement and / or separation, as well as by posting advertisements or articles in the media (social or conventional) in the French-speaking part of Switzerland.

DETAILED DESCRIPTION:
Internet-based self-help interventions have proved to have beneficial effects on a broad range of disorders including complicated grief disorder. Additionally, initial evidence is provided for the effectiveness of a cognitive-behaviorally-oriented online guided intervention for the milder grief symptoms. Unguided online interventions have a favorable cost-benefit ratio . French empirically supported online interventions are scarce, and to our knowledge, no such intervention exists for grieving individuals.

The primary purpose of this study is to evaluate the efficacy of this unguided internet-based self-help intervention on distress and well-being.

The secondary purpose is to assess the effects of the intervention on coping abilities, social integration and physical health after romantic bereavement or separation/divorce in adults. Additionally, the aim is to collect information about the users' perception of the program and their satisfaction with it. This information will be taken into account in order to develop an enhanced version of the program.

The primary outcomes are: distress symptoms (grief, depression, and anxiety) and well-being (satisfaction with life and eudaimonic well-being).

The main secondary outcomes are: coping abilities (grief-related avoidance, coping style), social integration (loneliness and social support), and finally the physical health state (physical symptoms and sleep quality).

Additionally, information about the satisfaction with the program will be collected and taken into account to develop a second, enhanced version of the program.

The design is a non-controlled evaluation pilot study with pre-, post- and follow-up assessments.

Participants fulfilling all the following inclusion criteria are eligible for the study:

* Romantic bereavement or separation/divorce. Either of these events must have happened more than 6 months before participating in the study.
* Subjective distress and need for support to cope with the loss
* Age: 20 years or older
* Regular internet access
* Mastery of the French language
* Approved Informed Consent (Appendix Informed Consent Form)

The presence of any of the following exclusion criteria will lead to exclusion of the participant :

* Moderate to acute current suicidality
* Severe psychological or somatic disorders which need immediate treatment.
* Concomitant psychotherapy (participants may take part in the self-help intervention, but will not be included in the study.)
* Prescribed drugs against depression or anxiety, if prescription or dosage has changed in the month prior or during the self-help intervention.
* Inability to follow the procedures of the study, e.g. due to comprehension problems
* Enrollment of the investigator, their family members, employees and other dependent persons.

Measurements: online-questionnaires will be used to assess the effects of the intervention at three measurement points: at baseline, at 12-weeks directly after the intervention and at follow-up 3-months after the end of the intervention.

Procedure: Participants will be recruited by contacting several grief-related associations in the French-speaking area of Switzerland, and by posting ads in the (social) media (see Appendices 9 and 10). First, interested persons will fill in a short questionnaire checking the participation criteria. Then, if eligible, they will approve the online informed consent and complete the baseline measures. Next, participants receive their login details for the internet-based self-help intervention. The 10 sessions will be self-administrated. The recommendation is to spend one week per session. Participants are free to go through the sessions as often as they wish.

The intervention is a non-controlled unguided internet-based self-help intervention for adults who seek support for coping with prolonged grief symptoms after romantic bereavement or separation/ divorce. The self-help program consists of 10 text-based sessions based on cognitive-behavioral psychotherapy techniques.

There will be no control intervention. However, the results (effect sizes) will be compared to the ones of the original authors of the program , who administered the same intervention to a German-speaking population (note however that the original program is an internet-based guided intervention, where weekly e-mail support was offered to the participants). The study will include at least 23 participants.

ELIGIBILITY:
Inclusion Criteria:

* Romantic bereavement or separation/divorce. Either of these events must have happened more than 6 months before participating in the study.
* Subjective distress and need for support to cope with the loss
* Age: 20 years or older
* Internet access
* Mastery of the French language
* Approved Informed Consent (Appendix Informed Consent Form)

Exclusion Criteria:

* Moderate to acute current suicidality (BDI-II item 9 > 1)
* Severe psychological or somatic disorders which need immediate treatment.
* Concomitant psychotherapy (participants may take part in the self-help intervention, but will not be included in the study.)
* Prescribed drugs against depression or anxiety, if prescription or dosage has changed in the month prior or during the self-help intervention.
* Inability to follow the procedures of the study, e.g. due to comprehension problems
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
Change in complicated grief symptoms (score at the Inventory of Complicated Grief) | Pretest / 12-week posttest / 3-month Follow-up
  assessed with: Inventory of Complicated Grief (Prigerson et al., 1995; Zech, 2012), on a scale ranging from 0 = never to 4 = always. The mean score is used as a final score. Higher score represent a higher symptom load.

SECONDARY OUTCOMES:
Change in Anxiety and Depression symptoms (score at the Hospital Anxiety and Depression Scale) | Pretest / 12-week posttest / 3-month Follow-up
  assessed with the Hospital Anxiety and Depression Scale (Savard, Laberge, Gauthier, Ivers, & Bergeron, 1998; Zigmond & Snaith, 1983). The mean score is used as a final score. Higher score represent a higher symptom load.
Change in Psychological Well-Being (score at the Psychological Well-Being Scales) | Pretest / 12-week posttest / 3-month Follow-up
  Psychological Well-Being Scales (Bouffard & Lapierre, 1997; Ryff, 1989; van Dierendonck, 2004) assessed on a scale ranging from 1 = I completely disagree, to 6 = I completely agree. The mean score is used as a final score. Higher score represent a better psychological well-being.
Change in Satisfaction with Life (score at the Satisfaction with Life Scale) | Pretest / 12-week posttest / 3-month Follow-up
  Satisfaction with Life Scale (Blais, Vallerand, Pelletier, & Brière, 1989; Diener, Emmons, Larsen, & Griffin, 1985) assessed on a scale ranging from 1 = I disagree strongly, to 7 = I agree strongly. The mean score is used as a final score. Higher score represent a better satisfaction with one's own life.
Change in Grief-Related Avoidance (score at the Grief-Related Avoidance Questionnaire) | Pretest / 12-week posttest / 3-month Follow-up
  Grief-Related Avoidance Questionnaire (Shear et al., 2007), assessed on a scale ranging from 0 = never to 4 = always. The mean score is used as a final score. Higher scores represent a higher tendency to avoid situations that could remind of the loss and is associated with worse outcomes.
Change in Coping strategies (score at the Brief-COPE) | Pretest / 12-week posttest / 3-month Follow-up
  Brief-COPE (Carver, Scheier, & Weintraub, 1989; Muller & Spitz, 2003) assesses 14 different typical coping strategies (Active coping, Planning, Suppression of competing activities, Restraint coping, Seeking social support - instrumental, Seeking social support - emotional, Positive reinterpretation & growth, Acceptance, Turning to religion, Focus on & venting of emotions, Denial, Behavioral disengagement, Mental disengagement, Alcohol-drug disengagement) on a scale ranging from 1 = not at all, to 4 = always. The average of each dimension is used separately. Higher scores represent a higher use of the coping strategy.
Change in loneliness (score at the De Jong Gierveld Short Scale for Emotional and Social Loneliness, short version) | Pretest / 12-week posttest / 3-month Follow-up
  Short Version of the De Jong Gierveld Short Scale for Emotional and Social Loneliness (de Jong Gierveld & van Tilburg, 2010; Vandenbroucke et al, 2012), on a scale ranging from 1 = yes, to 3 = no. The mean score is used as a final score. Higher score represent a higher self-perceived loneliness.
Change in perceived social support (score at the Social Support Questionnaire) | Pretest / 12-week posttest / 3-month Follow-up
  Social Support Questionnaire (Bruchon-Schweitzer, Rascle, Gelie, Fortier, Sifakis, & Constant, 2003; Sarason, Sarason, Shearin, & Pierce, 1987) on a scale ranging from 1 = very unsatisfied, to 6 = very satisfied. The mean score is used as a final score. Higher scores represent a higher satisfaction with the available social support.
Change in sleep problems (score at the Pittsburgh Sleep Quality Index) | Pretest / 12-week posttest / 3-month Follow-up
  The Pittsburgh Sleep Quality Index (PSQI; Blais, Gendron, Mimeault, & Morin, 1997; Buysse, Reynolds, Monk, Berman, & Kupfer, 1989) includes 19 self-rated questions about a variety of factors relating to sleep quality. They are then grouped into 7 components scores, each weighted equally on a 0-3 scale. These scores are then summed in a global PSQI score (range 0-21). A higher score represents more sleep problems.
Change in physical symptoms (score at the Physical Health Questionnaire) | Pretest / 12-week posttest / 3-month Follow-up
  The Physical Health Questionnaire (Kroenke, Spitzer, & Williams, 2002; Maggiori, 2010) assesses 15 physical symptoms on a scale ranging from 1 = not at all bothered, to 3 = very much bothered. The mean score is used as a final score. Higher scores represent a higher symptom load.
Satisfaction with the program (utility, clarity, impact, etc.) | 12-week Posttest
  Self-designed questionnaire assessing different quantitative and qualitative questions on the satisfaction with the program. These questions will be evaluated separately.

CONTACTS AND LOCATIONS:
Overall Officials: Valentino Pomini, Prof., Study Director — University of Lausanne
Locations (1):
- University of Lausanne - Institute of Psychology, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
After publishing the results, we will make the codified data available on request.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Access Criteria: We demand that the purpose of the request is clearly stated.

REFERENCES:
- [Background] Efinger, L., Debrot, A., & Pomini, V. (2021). LIVIA-FR : Implémentation et évaluation d'une intervention par Internet pour des personnes francophones peinant à surmonter la perte de leur partenaire. Annales Médico-Psychologiques, Revue Psychiatrique. Advance online publication. https://doi.org/10.1016/j.amp.2021.05.004
- See also: Recruitment page — http://www.psyconsultonline.ch